CLINICAL TRIAL: NCT04007588
Title: A Phase II Trial of Neoadjuvant Treatment With PD-1 Inhibition (Nivolumab) With or Without IDO Inhibition (BMS-986205) and With or Without CTLA-4 Inhibition (Ipilimumab) in Resectable Stage III or IV Melanoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Elizabeth Buchbinder, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19-043
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Melanoma Stage III; Melanoma Stage IV
Keywords: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Nivolumab; linrodostat; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Nivolumab+BMS-986205 (Experimental): * Nivolumab will be administered intravenously Day 1 of each 28 day cycle.
  * BMS-986205 will be administered orally on a daily basis
  Interventions: Drug: Nivolumab; Drug: BMS-986205
- Nivolumab (Experimental): -Nivolumab will be administered intravenously Day 1 of each 28 day cycle.
  Interventions: Drug: Nivolumab
- Nivolumab+Ipilimumab (Experimental): * Nivolumab will be administered intravenously Day 1 of each 28 day cycle.
  * Ipilimumab will be administered intravenously every 6 weeks
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — Nivolumab is a types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells. Nivolumab work by stopping various molecules on cancer cells and body cells from working against the immune system's natural fight against cancer
  Other Names: OPDIVO
Drug: BMS-986205 — BMS-986205 is a types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells. BMS-986205 work by stopping various molecules on cancer cells and body cells from working against the immune system's natural fight against cancer
  Arms: Nivolumab+BMS-986205
Drug: Ipilimumab — Ipilimumab is a types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells. Ipilimumab work by stopping various molecules on cancer cells and body cells from working against the immune system's natural fight against cancer
  Other Names: YERVOY
  Arms: Nivolumab+Ipilimumab

SUMMARY:
This research study is studying different immunotherapy regimens as a possible treatment for stage III or IV resectable melanoma.

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug to learn whether the drug works in treating a specific disease. "Investigational" means the drug is being studied.

The FDA (the U.S. Food and Drug Administration) has approved OPDIVO® (nivolumab), YERVOY® (ipilimumab), and a combination of the two as treatment options for metastatic melanoma.

The FDA (the U.S. Food and Drug Administration) has not approved the combination of nivolumab and BMS-986205 as a treatment for any disease. This research study is looking for more information on the efficacy the combination of nivolumab and BMS-986205 in the treatment of melanoma.

Nivolumab, Ipilimumab, and BMS-986205 are types of immunotherapy. Immunotherapy works by encouraging the body's own immune system to attack the cancer cells. Nivolumab, Ipilimumab, and BMS-986205 work by stopping various molecules on cancer cells and body cells from working against the immune system's natural fight against cancer.

In this research study, the investigators are going to look at the following while the participants are receiving the study drug(s):

• The effectiveness (how well the drug works), safety, and tolerability of Nivolumab, BMS-986205 and Nivolumab, and Ipilimumab and Nivolumab in people with resectable stage III or IV melanoma

ELIGIBILITY:
Inclusion Criteria:

* Histologic or cytologic diagnosis of resectable stage III or IV cutaneous melanoma. Patients with melanoma of mucosal origin are not eligible. Patients with acral melanoma that fit criteria are eligible. Patients must have clinically detectable stage III (clinically detectable N1b, N1c, N2b, N2c, N3b or N3c) or stage IV resectable melanoma.
* Age ≥ 18 years.
* ECOG performance status ≤2 (Karnofsky ≥60%, see Appendix A)
* Participants must have normal organ and marrow function as defined below:

  * leukocytes ≥2,000/mcL
  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥9.0g/dL
  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * creatinine within normal institutional limits OR
  * creatinine clearance ≥40 mL/min/1.73 m2 for participants with creatinine levels above institutional normal.
  * C-Reactive Protein < institutional ULN
* Quantitative or qualitative G6PD assay results must not suggest underlying G6PD deficiency
* Measurable disease (by CT, PET/CT or MRI)
* Prior therapies including targeted therapy and immunotherapy are not allowed, with the exception of adjuvant Ipilimumab or Interferon-α-2b.
* Ability to understand and the willingness to sign a written informed consent document.
* Ability to swallow pills intact and without GI issues which may impact medication absorption.
* Women of childbearing potential (WOCBP) must agree to follow instructions for method(s) of contraception (Refer to Appendix B) for the duration of treatment with study treatment(s) plus 5 months post-treatment completion (i.e. 30 days plus the time required for nivolumab to undergo approximately 5 half-lives).
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study treatment.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study treatment(s) plus 7 months post-treatment completion (i.e. 90 days plus the time required for nivolumab to undergo approximately 5 half-lives). In addition, male participants must be willing to refrain from sperm donation during this time. This criterion applies to azoospermic males as well.

Exclusion Criteria:

* A history of prior treatment with PD-1 inhibitor, CTLA-4 inhibitor or IDO inhibition. Prior therapy with ipilimumab or Interferon-α-2b in the adjuvant setting is permitted. Participants may not have received live/attenuated vaccines within 30 days of first treatment.
* Participants with uveal or mucosal melanoma
* Participants with known brain metastases must have documented stability for at least 30 days directly prior to study enrollment and not be requiring active treatment for these. Prior radiation, surgery and stereotactic radiosurgery are allowed but must be completed four weeks prior to initiating therapy.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to nivolumab, ipilimumab, methylene blue or BMS-986205. History or presence of hypersensitivity or idiosyncratic reaction to methylene blue.
* Need for systemic steroids at the time of enrollment. Physiologic replacements at a dose of less than 10 mg daily prednisone equivalent is allowed.
* Blood Methemoglobin > ULN, assessed in an arterial or venous blood sample or by co-oximetry
* Participants with active ILD/pneumonitis or history of ILD/ pneumonitis requiring steroids.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab or BMS-986205, breastfeeding should be discontinued if the mother is treated with nivolumab or BMS-986205. These potential risks may also apply to other agents used in this study.
* Known active HIV, Hepatitis B or Hepatitis C patients. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for an immunologic effect with the therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Autoimmune disease that requires treatment at the time of enrollment. Participants with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic treatment or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Participant with a personal or family (ie, in a first-degree relative) history of cytochrome b5 reductase deficiency (previously called methemoglobin reductase deficiency) or other diseases that put them at risk of methemoglobinemia. All participants will be screened for methemoglobin levels prior to randomization.
* Participant with a history of G6PD deficiency or other congenital or autoimmune hemolytic disorders. All participants will be screened for G6PD levels prior to randomization.
* Participants must not have a history of life-threatening toxicity related to prior immune therapy (eg. anti-CTLA-4 or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways) except those that are unlikely to re-occur with standard countermeasures (eg. hormone replacement after adrenal crisis).
* Treatment with botanical preparations (eg, herbal supplements or traditional Chinese medicines) intended for general health support or to treat the disease under study within 2 weeks prior to randomization.
* History of other malignancy within 3 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of > 90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or Stage I uterine cancer.
* Participants who have had major surgery requiring general anesthesia or significant trauma who have not recovered per physician determination for at least 14 days prior to randomization.
* Participants with conditions known to interfere significantly with the absorption of oral medication, as per investigator judgment.
* Participants with uncontrolled adrenal insufficiency.
* Prior history of serotonin syndrome.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-06 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Major Pathologic Response Rate | 2 years
  Complete Pathological response rate or near pathological complete response rate on each treatment arm

SECONDARY OUTCOMES:
Recurrence free survival | 2 years
  Time from treatment start to recurrence of melanoma
Overall Survival Rate | 2 years
  Time from treatment start to death
Changes In Infiltrating immune cells From Pre-Treatment To Time Of Excision | 2 Years
  Changes in immune cells in the tumor micro environment including CD8 T-cells
Rates of adverse events and serious adverse events on the different treatment arms. | 2 years
  Rates of different grade adverse events on each treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth I Buchbinder, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BCH - Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu BIDMC - Contact the Beth Israel Deaconess Medical Center Technology Ventures Office at tvo@bidmc.harvard.edu BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu MGH - Contact the Partners Innovations team at http://www.partners.org/innovation